CLINICAL TRIAL: NCT00686751
Title: Immunomodulatory Effects of Vitamin D in Chronic Hemodialysis Patients
Brief Title: Immune Effects of Vitamin D in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renal Research Institute (Other)
Collaborators: Abbott (Industry)
Responsible Party: Nathan Levin, MD, Renal Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 223-04
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: End Stage Renal Disease; Hemodialysis; Inflammatory Response; Cardiovascular Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): There is only one arm in this study. Each subject will be studied through 3 phases lasting a total of 4 weeks:
  Phase 1: administration of study medication at the end of hemodialysis treatment.
  Phase 2: no administration of study medication. Phase 3: administration of study medication at the beginning of hemodialysis.
  Interventions: Drug: paricalcitol

INTERVENTIONS:
Drug: paricalcitol — Dosage Form: Intravenous administration. Dosage: 0.01 micrograms/kilogram of body weight. Frequency: 2 HD treatments of each study week (depending on phase of study). Duration: 4 weeks.

SUMMARY:
The purpose of this study to examine whether vitamin D can reduce the activation of the immune system during dialysis. When activated, the immune cells release certain substances, called cytokines, which can be measured from small blood samples. We want to study to what degree the immune system is activated during a regular dialysis treatment and whether the time point of vitamin D administration, either right before the start or right at the end of a dialysis treatment, has an impact on the activation of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Patient stable on chronic hemodialysis for more than 3 months.
* PTH level between 150 - 800 pg/ml.
* Ability to give informed consent.
* Serum calcium levels (corrected for albumin level of 4.0 g/dL) less than 10.5 mg/dL for the last three consecutive measurements.
* Serum Phosphorus levels between 2.5 and 7.0 mg/dL for the last three consecutive measurements.
* Ca x P-Product of less than 75 mg2/dL2 in the last three consecutive measurements.

Exclusion Criteria:

* Known active malignancy.
* Liver disease defined as serum aspartate aminotransferase, alanine aminotransferase, or gamma-glutamyltransferase levels more than 2 times the upper limits of normal.
* PTH levels between 150 pg/mL and 800 pg/mL.
* Hypercalcemia or hypercalcemic episodes within the last 4 weeks.
* Ca x P-Product more than 75 mg2/dL2 within the last 4 weeks.
* Any clinical significant infections which are or have been treated with antibiotics within 6 weeks prior to start of the study.
* Chronic viral infection (HIV, Hepatitis B or C).
* Currently on immunosuppressive medication (steroids, cyclosporine, etc…).
* Hematocrit less than 30 %.
* History of blood disorders other than renal anemia.
* Age of less than 18 years or more than 75 years.
* Hypersensitivity to paricalcitol or any ingredient of the product.
* Parathyroidectomy.
* Participation in another study at the same time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
measurement of pro- and anti-inflammatory cytokines and inflammatory markers | first and second HD treatments for the 4 weeks of the study

SECONDARY OUTCOMES:
serum calcium level | 24 hours after termination of second HD treatment in week 3 of study
serum phosphate level | 24 hours after termination of second HD treatment in week 3 of study

CONTACTS AND LOCATIONS:
Overall Officials: Nathan W Levin, MD, Principal Investigator — Renal Research Institute
Locations (3):
- United States (3):
  - Irving Place Dialysis Center, New York, New York
  - Upper Manhattan Dialysis Center, New York, New York
  - Yorkville Dialysis Center, New York, New York